CLINICAL TRIAL: NCT00550745
Title: A Phase IV Clinical Trial to Evaluate the Safety and Tolerability of ZOSTAVAX™ in Subjects ≥ 60 Years of Age
Brief Title: ZOSTAVAX™ Safety Study in Subjects ≥ 60 Years of Age (V211-020)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V211-020; 2007_606
Record Dates: First submitted 2007-10-29; First posted 2007-10-30 (Estimated); Results first posted 2010-02-02 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-03

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Arm 1: vaccine
  Interventions: Biological: Zoster Vaccine, Live
- 2 (Placebo Comparator): Arm 2: Placebo Comparator
  Interventions: Biological: Comparator: placebo

INTERVENTIONS:
Biological: Zoster Vaccine, Live — single 0.65 mL Zoster Vaccine, Live injection. 6 month treatment period.
  Arms: 1
Biological: Comparator: placebo — single 0.65 mL Placebo injection. 6 month treatment period.
  Arms: 2

SUMMARY:
The purpose of the study is to evaluate the general safety of ZOSTAVAX™ in subjects 60 years of age or older as required by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* 60+ years of Age
* Signed an informed consent prior to the start of study
* Non-Feverish, (less than 101.0°F / 38.3°C) on day of vaccination
* Females must be postmenopausal or have a negative pregnancy test

Exclusion Criteria:

* A history of allergic reaction to any vaccine component (including gelatin or neomycin)
* Prior receipt of any varicella or zoster vaccine
* Any live virus vaccine administered within 4 weeks before the start of the study or scheduled during the 42 days after vaccination
* Any inactivated virus vaccine, except for flu vaccine, administered within 7 days before the start of the study or scheduled during the 42 days after vaccination
* Subject is pregnant or breastfeeding
* Participation in an investigational drug or vaccine study within the last 30 days prior to the start of the study or expected during the 42 days after vaccination
* An ongoing illness (including active untreated tuberculosis) that might interfere with or prevent the subject from completion of the study
* Use of immunosuppressive therapy. Subjects taking corticosteroids such as prednisone should be excluded. Excluded immunosuppressive therapies also include chemotherapeutic agents used to treat cancer or other conditions, and treatments associated with organ or bone marrow transplantation
* Known or suspected immune dysfunction that is caused by a medical condition or any other cause. Examples of medical conditions associated with immune dysfunction include congenital immunodeficiency, human immunodeficiency virus (HIV) infection, organ or bone marrow transplantation, leukemia, lymphoma, Hodgkin's disease, multiple myeloma, or generalized malignancy. Subjects with a history of cancer who are not on active treatment and are not thought to have a weakened immune system at the time of enrollment will be eligible
* Any active use of non-topical antiviral therapy including but not limited to acyclovir, famciclovir, valacyclovir, ganciclovir, foscarnet, brivudine, and cidofovir

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11999 (Actual)
Dates: Start 2007-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Murray AV, Reisinger KS, Kerzner B, Stek JE, Sausser TA, Xu J, Wang WW, Chan IS, Annunziato PW, Parrino J. Safety and tolerability of zoster vaccine in adults >/=60 years old. Hum Vaccin. 2011 Nov;7(11):1130-6. doi: 10.4161/hv.7.11.17982. Epub 2011 Nov 1. PMID 22048110

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase IV
  First subject enrolled on 17-Sep-2007.
  Last subject enrolled on 19-Jun-2008.
  The last subject's last visit was 15-Jan-2009.
  The study was conducted at 46 study centers throughout the United States, Canada, Germany,
  Spain, and United Kingdom.
Groups:
- ZOSTAVAX™; Placebo: Represents the number of randomized subjects according to the vaccination group as they were assigned at study entry and not the treatment, ZOSTAVAX™ or placebo, received.
Period: Overall Study
Arm/Group | ZOSTAVAX™ | Placebo
Started | 6000 | 5999
Completed | 5913 | 5939
Not Completed | 87 | 60
Not completed — Death | 20 | 16
Not completed — Lost to Follow-up | 45 | 30
Not completed — Physician Decision | 0 | 2
Not completed — Protocol Violation | 4 | 2
Not completed — Withdrawal by Subject | 17 | 10
Not completed — Screen failure | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- ZOSTAVAX™: Represents the number of subjects according to the treatment (ZOSTAVAX™) received.
  Excludes subjects who were not vaccinated.
- Placebo: Represents the number of subjects according to the treatment (placebo) received.
  Excludes subjects who were not vaccinated.
- Total: Total of all reporting groups
Arm/Group | ZOSTAVAX™ | Placebo | Total
Number analyzed (Participants) | 5983 | 5997 | 11980
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (7.5) | 70.4 (7.6) | 70.5 (7.5)
Age, Customized [Number; unit: participants] — Age Group (years)
  participants
    60 to 69 Years of Age | 3092 | 3113 | 6205
    70 to 79 Years of Age | 1994 | 1986 | 3980
    ≥ 80 Years of Age | 897 | 898 | 1795
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3515 | 3525 | 7040
  Male | 2468 | 2472 | 4940
Race/Ethnicity, Customized [Number; unit: participants]
  Black | 109 | 85 | 194
  White | 5759 | 5770 | 11529
  Other | 115 | 142 | 257
Region [Number; unit: Participants]
  U.S. | 5309 | 5312 | 10621
  Non-U.S. | 674 | 685 | 1359
Type of Residence [Number; unit: Participants]
  Assisted Living | 176 | 162 | 338
  Independent Residential | 5790 | 5821 | 11611
  Nursing Home | 17 | 14 | 31

OUTCOME MEASURES:

1. Primary Outcome: Serious Adverse Events Reported Within 42 Days Postvaccination
Description: Only Serious Adverse Events were collected and analyzed for this
  study.
  A serious adverse event is any adverse event that results in death, is life threatening, results in a persistent or significant disability/incapacity, results in hospitalization or prolongs an existing hospitalization, is a congenital anomaly/birth defect, is a cancer, is an overdose, or is considered an "other important medical event" based on medical judgement.
Time Frame: 42 Days
Population: All subjects who were vaccinated according to actual treatment received (ZOSTAVAX™ or placebo) and had safety follow-up.
  Death - Number of subjects that had a fatal serious adverse event with an onset date within the 42 day reporting period. The date of death may have occurred after 42 days.
Measure: Number; unit: Participants
Groups:
- ZOSTAVAX™: All subjects who were vaccinated according to actual treatment received (ZOSTAVAX™) and had safety follow-up.
- Placebo: All subjects who were vaccinated according to actual treatment received (Placebo) and had safety follow-up.
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 5979 | 5990
Participants
  Serious Adverse Events (AEs) | 84 | 67
  Serious AEs deemed vaccine-related by investigator | 2 | 0
  Death | 6 | 5
Statistical Analysis 1: Comparison: ZOSTAVAX™ vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.26, 95% CI [0.91 to 1.73] — Relative risk (ZOSTAVAX™/placebo) of proportion of subjects reporting ≥ 1 serious AE through 42 Days postvaccination and 95% Confidence Interval were based on Miettinen and Nurminen [Comparative analysis of two rates. Stat Med 1985;4:213-26] method

2. Secondary Outcome: Serious Adverse Events Reported Within 6 Months (Day 1 to 182) Postvaccination
Description: as for outcome 1
Time Frame: 6 months
Population: All subjects who were vaccinated according to actual treatment received (ZOSTAVAX™ or placebo) and had safety follow-up.
  Death - Number of subjects that had a fatal serious adverse event with an onset date within the 182 day reporting period. The date of death may have occurred after 182 days.
Measure: Number; unit: Participants
Arm/Group | ZOSTAVAX™ | Placebo
Number analyzed (Participants) | 5979 | 5990
Participants
  Serious AEs | 340 | 300
  Serious AEs deemed vaccine-related by investigator | 2 | 1
  Death | 24 | 17
Statistical Analysis 1: Comparison: ZOSTAVAX™ vs Placebo; Test type: Superiority or Other; Risk Ratio (RR) = 1.13, 95% CI [0.98 to 1.32] — Relative risk (ZOSTAVAX™/placebo) of proportion of subjects reporting ≥ 1 serious AE through 6 months postvaccination and 95% Confidence Interval were based on Miettinen and Nurminen [Comparative analysis of two rates. Stat Med 1985;4:213-26] method

ADVERSE EVENTS:
Time Frame: Serious AEs reported within 6 months (182 days) postvaccination. Only Serious adverse events were collected in this study. The "Other Adverse Events" table is not applicable for this study and shows "0/0" for " participants affected/at risk"
Description: Subjects were instructed to call the site immediately, at any time during the study, if they experienced a serious adverse event. Subjects were also called by study staff at 42 days, 4 months, and 6 months postvaccination, using a prespecified phone script, to determine if subjects had a previously unreported serious adverse event.
Arm/Group | ZOSTAVAX™ | Placebo
Serious Adverse Events (participants affected / at risk) | 340/5979 | 300/5990
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ZOSTAVAX™ (N=5979) | Placebo (N=5990)
Anaemia (Blood and lymphatic system disorders) | 4 | 2
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 | 1
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Macrocytosis (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 4 | 0
Acute myocardial infarction (Cardiac disorders) | 3 | 2
Angina pectoris (Cardiac disorders) | 0 | 3
Angina unstable (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 1 | 2
Atrial fibrillation (Cardiac disorders) | 21 | 14
Atrial flutter (Cardiac disorders) | 5 | 0
Atrioventricular block (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 6 | 2
Bundle branch block right (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac disorder (Cardiac disorders) | 2 | 0
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 8 | 9
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 11 | 15
Coronary artery occlusion (Cardiac disorders) | 0 | 1
Coronary artery restenosis (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Mitral valve prolapse (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 8 | 14
Myocardial ischaemia (Cardiac disorders) | 1 | 1
Palpitations (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 2 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 2
Ventricular extrasystoles (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular hypertrophy (Cardiac disorders) | 1 | 0
Wandering pacemaker (Cardiac disorders) | 0 | 1
Arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Meniere's disease (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 1 | 0
Hyperaldosteronism (Endocrine disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 1
Uveitis (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal mass (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Appendicitis perforated (Gastrointestinal disorders) | 1 | 1
Colitis (Gastrointestinal disorders) | 2 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 1 | 0
Colonic polyp (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Gastroduodenitis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 7 | 2
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Hiatus hernia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 2 | 0
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 | 0
Intestinal fistula (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 2 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 4
Pancreatitis acute (Gastrointestinal disorders) | 4 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Adhesion (General disorders) | 1 | 0
Catheter related complication (General disorders) | 1 | 0
Chest discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 12 | 17
Death (General disorders) | 2 | 1
Hernia obstructive (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 5 | 2
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 2
Cholecystitis acute (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 1
Abdominal abscess (Infections and infestations) | 2 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Bone abscess (Infections and infestations) | 0 | 1
Bronchiectasis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 3
Cellulitis (Infections and infestations) | 1 | 8
Cholecystitis infective (Infections and infestations) | 1 | 0
Clostridial infection (Infections and infestations) | 1 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 8 | 4
Empyema (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 5 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 3
Herpes zoster (Infections and infestations) | 0 | 2
Lemierre syndrome (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 2 | 3
Meningitis (Infections and infestations) | 0 | 1
Meningitis aseptic (Infections and infestations) | 1 | 0
Necrotising fasciitis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 0 | 1
Pleural infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 16 | 13
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 0 | 1
Post procedural infection (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 2
Pseudomembranous colitis (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 2 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 6 | 1
Septic phlebitis (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 3
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 0 | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic complication (Injury, poisoning and procedural complications) | 1 | 0
Anastomotic stenosis (Injury, poisoning and procedural complications) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0
Coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Dislocation of joint prosthesis (Injury, poisoning and procedural complications) | 0 | 2
Eyeball rupture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Foreign body trauma (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 1
Graft thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 3
Implantable defibrillator malfunction (Injury, poisoning and procedural complications) | 1 | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 | 1
Incision site haematoma (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Patella fracture (Injury, poisoning and procedural complications) | 2 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 5
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Thrombosis in device (Injury, poisoning and procedural complications) | 0 | 2
Tracheal injury (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Blood glucose increased (Investigations) | 0 | 1
Blood sodium decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Arthrofibrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 4 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 14 | 10
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 | 2
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 12 | 7
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Breast cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Cardiac myxoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hodgkin's disease stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mycosis fungoides (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloma recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neurilemmoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian low malignant potential tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Peritoneal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 6
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 14 | 8
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid artery disease (Nervous system disorders) | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 2
Cerebellar infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 2 | 6
Convulsion (Nervous system disorders) | 2 | 0
Dementia (Nervous system disorders) | 1 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Global amnesia (Nervous system disorders) | 0 | 1
Intracranial aneurysm (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 1
Lumbar radiculopathy (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 1 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 2
Presyncope (Nervous system disorders) | 1 | 2
Radiculopathy (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 10 | 5
Syncope vasovagal (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 2 | 6
Affective disorder (Psychiatric disorders) | 1 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Catatonia (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 1
Dissociative identity disorder (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Acute prerenal failure (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 0 | 1
Hypotonic urinary bladder (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 3 | 0
Renal failure acute (Renal and urinary disorders) | 12 | 2
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 2
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 2
Epididymitis (Reproductive system and breast disorders) | 1 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Rectocele (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 11
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Thyroidectomy (Surgical and medical procedures) | 0 | 1
Accelerated hypertension (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 2 | 1
Aortic dissection (Vascular disorders) | 0 | 2
Aortic stenosis (Vascular disorders) | 1 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Femoral arterial stenosis (Vascular disorders) | 1 | 0
Femoral artery aneurysm (Vascular disorders) | 0 | 1
Haematoma (Vascular disorders) | 2 | 0
Hypertension (Vascular disorders) | 3 | 2
Hypotension (Vascular disorders) | 3 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Peripheral vascular disorder (Vascular disorders) | 2 | 0
Temporal arteritis (Vascular disorders) | 2 | 0
Vasculitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.